CLINICAL TRIAL: NCT03618550
Title: Phase II Study of Second-line Pembrolizumab Plus GVD for Relapsed or Refractory Hodgkin Lymphoma
Brief Title: Phase II Study of Second- Line Pembrolizumab Plus GVD for Relapsed or Refractory Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-160
Record Dates: First submitted 2018-07-30; First posted 2018-08-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin Lymphoma; Relapsed or Refractory Hodgkin Lymphoma
Keywords: Pembrolizumab; GVD; 18-160
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — pembrolizumab; Gemcitabine; Vinorelbine; liposomal doxorubicin; Hematopoietic Stem Cell Mobilization

STUDY DESIGN:
Intervention Model Description: This is a phase II study evaluating pembrolizumab plus gemcitabine, vinorelbine, liposomal doxorubicin (GVD) in transplant eligible patients with relapsed or refractory Hodgkin lymphoma following failure of 1-line of multi-agent chemotherapy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Safety Window and DLT definition (Part 1) (Experimental): Initially, 6 patients will be treated on the safety portion of the study and observed for dose limiting toxicities (DLTs). If 1 or fewer patients experience dose[1]limiting toxicity (DLT), enrollment onto the study will proceed according to a phase II, Simon 2- stage design.
  Interventions: Drug: pembrolizumab; Drug: gemcitabine; Drug: vinorelbine; Drug: liposomal doxorubicin; Procedure: Stem cell mobilization and collection
- Safety monitoring beyond after completion of safety window (PART 1) (Experimental): During the phase II portion of the study, patients will continue to be monitored for DLTs, adverse events, and events of interest throughout treatment with pembrolizumab-GVD, ASCT (part 1, if applicable), and 100 days following the last dose of pembrolizumab. Total planned enrollment is 39 patients
  Interventions: Drug: pembrolizumab; Drug: gemcitabine; Drug: vinorelbine; Drug: liposomal doxorubicin; Procedure: Stem cell mobilization and collection
- Autologous Stem Cell Transplant (ASCT) (PARTS 1 and 3) (Experimental): Stem cell mobilization and collection will be performed as per institutional guidelines after 2-4 cycles of pembrolizumab-GVD.
  Interventions: Drug: pembrolizumab; Drug: gemcitabine; Drug: vinorelbine; Drug: liposomal doxorubicin; Procedure: Stem cell mobilization and collection
- Pembrolizumab maintenance (PART 2) (Experimental): In part 2 of the study, patients who achieve complete response after 4 cycles of pembrolizumab[1]GVD will receive single-agent pembrolizumab for 13 cycles, which will begin 3-5 weeks after cycle 4 of pembrolizumab-GVD.
  Interventions: Drug: pembrolizumab; Drug: gemcitabine; Drug: vinorelbine; Drug: liposomal doxorubicin; Procedure: Stem cell mobilization and collection
- Pembrolizumab maintenance, third-line therapy, and HDT/ASCT (PART 3) (Experimental): In part 3 of the study, patients who achieve complete response after 2 cycles of pembrolizumab[1]GVD will be randomized to either consolidation with autologous stem cell transplant (after an additional optional 1-2 cycles of pembro-GVD) or 2 cycles of pembro-GVD followed by single agent pembrolizumab maintenance for 13 cycles.
  Interventions: Drug: pembrolizumab; Drug: gemcitabine; Drug: vinorelbine; Drug: liposomal doxorubicin; Procedure: Stem cell mobilization and collection
- Involved-site radiation therapy (ISRT) (PART 3) (Experimental): Patients with limited sites of disease prior to initiation of pembro-GVD are eligible to receive ISRT prior to ASCT with pembrolizumab maintenance.
  Interventions: Drug: pembrolizumab; Drug: gemcitabine; Drug: vinorelbine; Drug: liposomal doxorubicin; Procedure: Stem cell mobilization and collection

INTERVENTIONS:
Drug: pembrolizumab — Age 10-17: 2mg/kg (cap at 200mg), Age ≥ 18: 200 mg (flat) ,Day 1 of each 3 week cycle IV infusion 2-4 cycles (pre-ASCT)
Drug: gemcitabine — 1000mg/m^2 Days 1 and 8 of each 3 week cycle IV infusion 2-4 cycles
Drug: vinorelbine — 20mg/m^2 Days 1 and 8 of each 3 week cycle IV infusion 2-4 cycles
Drug: liposomal doxorubicin — 15mg/m^2 Days 1 and 8 of each 3 week cycle IV infusion 2-4 cycles
Procedure: Stem cell mobilization and collection — Stem cell mobilization and collection will be performed as per standard MSKCC guidelines after 2-4 cycles of pembrolizumab-GVD.

SUMMARY:
The purpose of this study is to test any good and bad effects of the study drug, pembrolizumab, in combination with GVD in the treatment of Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of classical Hodgkin's lymphoma. Primary refractory or relapsed disease proven by biopsy at enrolling institution.
* Stage I-III Hodgkin lymphoma (part 3)
* Relapse or refractory disease following 1 line of multi-agent chemotherapy (not including pembro-GVD).
* Eligible for HDT/ASCT
* Achieved complete response (Deauville 3 or better) per clinical review following 2 cycles of pembro-GVD
* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on Lugano 2014 criteria
* Have a performance status of 0 or 1 on the ECOG Performance Scale
* Demonstrate adequate organ function as defined in table below
* Demonstrate adequate organ function as defined in table below. Hematological*
* Absolute neutrophil count (ANC) ≥1000 /mcL
* Platelets ≥50,000 / mcL
* Hemoglobin ≥8 g/dL Renal
* Serum creatinine OR ≤1.5 X upper limit of normal (ULN) OR
* Measured or calculated creatinine clearance (eGFR can also be used in place of creatinine) ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic*
* Serum total bilirubin ≤ 1.5 X ULN OR ≤ 3 X ULN for subjects with liver metastases
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Pulmonary
* Hemoglobin-adjusted diffusing capacity for carbon monoxide ≥50% (If unadjusted DLCO is >/= 50% then there is no need to calculate adjusted) Cardiac
* Ejection fraction ≥45% Coagulation
* International normalized ratio (INR) OR prothrombin time (PT), Activated partial thromboplastin time (aPTT): ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

  *Lab values for eligibility should be based upon labs prior to Cycle 1 treatment of Pembro-GVD.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 2 weeks prior to receiving the first dose of study medication. On the day of planned treatment, if a blood pregnancy test has not been performed within the two week window, a stat pregnancy test (urine or blood) should be performed and the results reviewed before treatment is begun.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception (see details in section 11.4.3).
* Male subjects of childbearing potential must agree to use an adequate method of contraception.(see details in section 11.4.3).
* HIV-infected participants must have well-controlled HIV on ART, defined as:

  * Participants on ART must have a CD4+ T-cell count ≥350 cells/mm3 at the time of screening
  * Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening
  * It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months.
  * Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (Day 1) and agree to continue ART throughout the study
* Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible.

Exclusion Criteria:

* Received more than 1 prior treatment (combined modality therapy represents 1 treatment) for Hodgkin Lymphoma
* Known pregnancy or breast-feeding.

  * Breast-feeding should be discontinued prior to treatment initiation.
* Medical illness unrelated to Hodgkin's Lymphoma, which, in the opinion of the attending physician and/or principal investigator, makes participation in this study inappropriate.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known active HIV, Hepatitis B (e.g., Hepatitis B PCR positive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has not adequately recovered from major surgery or has ongoing surgical complications
* Has undergone solid organ transplant at any time, or prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Subjects who have had an allogeneic hematopoietic transplant greater than 5 years ago are eligible as long as there are no symptoms of GVHD.)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (part 1) | 2 years
  Response to pembrolizumab-GVD will be assessed using the RECIL criteria.

SECONDARY OUTCOMES:
Evaluate the 2-year PFS rate (part 2) | 2 years
  Only patients who receive the Pembrolizumab maintenance regime will be considered evaluable for 2-year PFS and OS rates.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - University of Miami, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Background] Moskowitz AJ, Shah G, Schoder H, Ganesan N, Drill E, Hancock H, Davey T, Perez L, Ryu S, Sohail S, Santarosa A, Galasso N, Neuman R, Liotta B, Blouin W, Kumar A, Lahoud O, Batlevi CL, Hamlin P, Straus DJ, Rodriguez-Rivera I, Owens C, Caron P, Intlekofer AM, Hamilton A, Horwitz SM, Falchi L, Joffe E, Johnson W, Lee C, Palomba ML, Noy A, Matasar MJ, Pongas G, Salles G, Vardhana S, Sanin BW, von Keudell G, Yahalom J, Dogan A, Zelenetz AD, Moskowitz CH. Phase II Trial of Pembrolizumab Plus Gemcitabine, Vinorelbine, and Liposomal Doxorubicin as Second-Line Therapy for Relapsed or Refractory Classical Hodgkin Lymphoma. J Clin Oncol. 2021 Oct 1;39(28):3109-3117. doi: 10.1200/JCO.21.01056. Epub 2021 Jun 25. PMID 34170745
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm